CLINICAL TRIAL: NCT01458951
Title: A Multicentre, Randomized, Double-blind, Placebo-controlled, Parallel-group Study Of Oral Cp-690,550 As An Induction Therapy In Subjects With Moderate To Severe Ulcerative Colitis.
Brief Title: A Study To Evaluate Both The Efficacy and Safety Profile of CP-690,550 In Patients With Moderately to Severely Active Ulcerative Colitis
Acronym: OCTAVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921095; 2011-004579-35 (EudraCT Number); OCTAVEINDUCTION2 (Other: Alias Study Number)
Record Dates: First submitted 2011-10-21; First posted 2011-10-25 (Estimated); Results first posted 2016-06-01 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-04

CONDITIONS: Ulcerative Colitis
Keywords: Tofacitinib; CP-690; 550; Moderate to severe ulcerative colitis; phase 3 clinical trial; Mayo score
MeSH Terms: conditions — Colitis, Ulcerative | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tofacitinib 10 mg BID (Experimental)
  Interventions: Drug: tofacitinib
- Placebo BID (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tofacitinib — 10 mg oral BID
  Other Names: CP-690,550
  Arms: tofacitinib 10 mg BID
Drug: Placebo — Placebo oral BID
  Arms: Placebo BID

SUMMARY:
This study is designed to evaluate the efficacy and safety of tofacitinib (CP-690,550) in patients with moderate to severe ulcerative colitis who have failed or be intolerant to one of following treatments for ulcerative colitis: oral steroids, azathiopurine/6-mercaptopurine, or anti-TNF-alpha therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age.
* Males and females with a documented diagnosis of UC at least 4 months prior to entry into the study.
* Subjects with moderately to severely active UC based on Mayo score criteria.
* Subjects must have failed or be intolerant of at least one of the following treatments for UC:

  * Corticosteroids (oral or intravenous).
  * Azathioprine or 6 mercaptopurine (6 MP).
  * Anti TNF therapy.

Exclusion Criteria:

* Presence of indeterminate colitis, microscopic colitis, ischemic colitis, infectious colitis, or clinical findings suggestive of Crohn's disease.
* Subjects with disease limited to distal 15 cm.
* Subjects without previous treatment for UC (ie, treatment naïve).
* Subjects displaying clinical signs of fulminant colitis or toxic megacolon.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 2012-06; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (182):
- United States (62):
  - Desert Sun Clinical Research, LLC, Tucson, Arizona
  - Desert Sun Gastroenterology, Tucson, Arizona
  - Desert Sun Surgery Center, Tucson, Arizona
  - Alliance Clinical Research, Oceanside, California
  - Clinical Application Laboratories, San Diego, California
  - San Diego Endoscopy Center, San Diego, California
  - UCSF Endoscopy Unit at Mount Zion, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - Bristol Hospital, Bristol, Connecticut
  - Connecticut Clinical Research Foundation, Bristol, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Central Connecticut Endoscopy Center, Plainville, Connecticut
  - Citrus Surgery & Endoscopy Center (Colonoscopy), Crystal River, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Suncoast Endoscopy Center (colonoscopy), Inverness, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Advanced Gastroenterology Center, Port Orange, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Endoscopy Center, Port Orange, Florida
  - Port Orange Urgent Care, Port Orange, Florida
  - Atlanta Center for Gastroenterology, P.C., Decatur, Georgia
  - Cotton-O'Neil Clinical Research Center, Digestive Health, Topeka, Kansas
  - Gastrointestinal Specialists, A.M.C., Shreveport, Louisiana
  - Shreveport Endoscopy Center, A.M.C., Shreveport, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Chevy Chase Endoscopy Center (Endoscopies Only), Chevy Chase, Maryland
  - MGG Group Co., Inc., Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Center for Digestive Health, Troy, Michigan
  - Surgical Centers of Michigan, Troy, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Surgery Center of Columbia, Columbia, Missouri
  - Hannibal Regional Hospital, Hannibal, Missouri
  - Audrain Medical Center, Mexico, Missouri
  - Center for Digestive & Liver Disease, Inc., Mexico, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - AGA Clinical Research Associates, LLC, Egg Harbor, New Jersey
  - South Jersey Gastroenterology, Marlton, New Jersey
  - The Gastroenterology Group of South Jersey, Vineland, New Jersey
  - The Endo Center at Voorhees, Voorhees Township, New Jersey
  - University of Rochester, Rochester, New York
  - Carolina Research - Carolina Digestive Diseases, Greenville, North Carolina
  - Regional Gastroenterology Associates of Lancaster, Ltd., Lancaster, Pennsylvania
  - Vanderbilt University Medical Center - IBD Clinic, Nashville, Tennessee
  - Vanderbilt University Medical Center - GI Research Office, Nashville, Tennessee
  - Vanderbilt University Medical Center - Drug Shipment, Nashville, Tennessee
  - Vanderbilt University Medical Center - GCRC, Nashville, Tennessee
  - Vanderbilt University Medical Center - Heart Station, Nashville, Tennessee
  - Vanderbilt University Medical Center - Radiology, Nashville, Tennessee
  - Texas Clinical Research Institiute, Arlington, Texas
  - Austin Gastroenterology PA/Professional Quality Research, Inc., Austin, Texas
  - Austin Gastroenterology PA, Austin, Texas
  - Austin Endoscopy Center II, Austin, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Digestive Health Specialists of Tyler, Tyler, Texas
  - VCU Health System Digestive Health Center, Richmond, Virginia
  - VCU Health System Endoscopy Suite, Richmond, Virginia
  - VCU Medical Center Investigational Drug Service (IDS), Richmond, Virginia
  - Virginia Commonwealth University, Clinical Research Services (CRSU), Richmond, Virginia
- Australia (5):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Concord Hospital -Concord Repatriation Hospital, Concord, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Liverpool Hospital Eastern Campus, Liverpool, New South Wales
  - Monash Medical Centre, Clayton, Victoria
- Austria (2):
  - Medizinische Universitat Innsbruck, Innsbruck
  - Krankenhaus Barmherzige Brueder St. Veit/Glan, Sankt Veit an der Glan
- Belgium (3):
  - GZA St Vincentius, Antwerp
  - AZ Groeninge, Campus Kennedylaan, Kortrijk
  - H-Hartziekenhuis Roeselare-Menen vzw, Roeselare
- Hospital de Clinicas de Porto Alegre - HCPA, Porto Alegre, Rio Grande do Sul, Brazil
- Canada (5):
  - University of Alberta Hospital - Walter C. Mackenzie Health Sciences Centre, Edmonton, Alberta
  - University of Alberta - Zeidler Ledcor Centre, Edmonton, Alberta
  - Montreal General Hospital - McGill University Health Centre, Montreal, Quebec
  - Saskatoon City Hospital, Saskatoon, Saskatchewan
  - Royal University Hospital, Saskatoon, Saskatchewan
- Instituto de Coloproctologia ICO S.A.S., Medellín, Antioquia, Colombia
- Croatia (3):
  - University Hospital Center Osijek, Clinic of Internal Medicine,, Osijek
  - University Hospital Center Rijeka, Rijeka
  - University Hospital Center Zagreb,Department of Gastroenterology, Zagreb
- Czechia (2):
  - Nemocnice Strakonice, a.s., Interni oddeleni, Strakonice
  - Krajska Zdravotni a.s., Masarykova nemocnice Usti nad Labem, o.z., Ústí nad Labem
- Denmark (3):
  - Bispebjerg Hospital, Copenhagen, NV
  - Hvidovre University Hospital, Hvidovre
  - Odense University Hospital, Odense C
- Estonia (8):
  - ECG Unit, Innomedica OU and Qualitas AS (ECG Only), Tallinn
  - Innomedica OU, Tallinn
  - X-Ray Unit, Qualitas AS (X-Ray Only), Tallinn
  - East Tallinn Central Hospital Internal Medicine Clinic, Tallinn
  - ECG Unit, East Tallinn Central Hospital, Tallinn
  - X-Ray Unit, East Tallinn Central Hospital, Tallinn
  - Quattromed HTI Laboratorid OU, Tallinn
  - Mammograaf OU (Endoscopy Only), Tallinn
- France (6):
  - Hopital Saint Andre, Bordeaux, France
  - CHU Amiens PICARDIE - Hopital SUD, Amiens
  - Hopital Beaujon, Clichy
  - Hopital Saint Antoine, Paris
  - C.H.U. de Reims - Hôpital Robert Debré, Reims
  - Hopital Nord, Saint-Priest-en-Jarez
- Germany (5):
  - Universitäetsklinik Schleswig-Holstein, Campus Kiel, Kiel, Schlewig Holstein
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt
  - Gastroenterologische Gemeinschaftspraxis Minden, Minden
  - University Hospital Munich-Grosshadern, Munich
  - Universitaetsklinikum Ulm, Ulm
- Hungary (9):
  - Dr. Rethy Pal Korhaz-Rendelointezet- III. Belgyogyaszat, Békéscsaba, Europe
  - Szent Janos Korhaz és Eszak-budai Egyesített Korhazak I Belgyogyaszat-Gasztroenterologiai Osztaly, Budapest
  - Peterfy Sandor utcai Korhaz- Rendelointezet es Baleseti Kozpontl. Belgyogyaszat, Budapest
  - MH Honvedkorhaz, Budapest
  - Pannonia Maganorvosi Centrum Kft., Budapest
  - Debreceni Egyetem Klinikai Központ Belgyógyászati Intézet, Gasztroenterológiai Tanszék, Debrecen
  - Bekes Megyei Pandy Kalman Korhaz, Gyula
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - "Karolina Korhaz Rendelointezet,Belgyogyaszat, Mosonmagyaróvár
- Israel (3):
  - Rambam Health Care Campus, Haifa
  - The Edith Wolfson Medical Center/Gastroenterology Institute, Holon
  - Kaplan Medical Center, Rehovot
- Daugavpils Regional Hospital, Daugavpils, Latvia
- Netherlands (3):
  - VU University Medical Center (VUMC), Amsterdam
  - Academic Medical Centre (AMC),, Amsterdam
  - University Medical Center Groningen (UMCG), Groningen
- New Zealand (6):
  - Christchurch Hospital, Christchurch, Canterbury
  - Auckland City Hospital, Auckland
  - Waikato Hospital, Hamilton
  - P3 Research Limited, Wellington
  - Pacific Radiology (X-rays only), Wellington
  - Bowen Hospital, Wellington
- Poland (7):
  - Centrum Medyczne Szpital Sw. Rodziny Sp. z o. o., Lodz, Iodzkie
  - Centrum Endoskopii Zabiegowej, Poradnia Chorob Jelitowych,, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Oddzial Chorob Wewnetrznych i Gastroenterologii,, Bialystok, Podlaskie Voivodeship
  - H-T Centrum Medyczne sp. z o.o. sp. komandytowa, Tychy, Silesian Voivodeship
  - Gabinet Endoskopii Przewodu Pokarmowego, Krakow
  - Endoskopia Sp. z.o.o., Sopot
  - Nzoz Vivamed, Warsaw
- Romania (2):
  - Spitalul Universitar de Urgenta Bucuresti, Sectia de Medicina Interna 2 si Gastroenterologie, Bucharest, Sector 5
  - Spitalul Clinic Judetean Mures, Sectia Clinica de Gastroenterologie, Jud. Mures
- Russia (8):
  - State budget institution of healthcare "City Clinical Hospital # 51 healthcare department of Moscow", Moscow, Russia
  - Municipal institution of healthcare "Clinical Hospital # 2", Yaroslavl, Russia
  - OOO Medical Center of Diagnostics and Prophylaxis "Sodruzhestvo", Yaroslavl, Russia
  - Federal state budget institution "State scientific centre of coloproctology", Moscow
  - State budget Healthcare Institution Moscow regional scientific research clinical institute, Moscow
  - Federal State Budgetary Institution "Scientific Research Institute of Physiology and, Novosibirsk
  - Municipal institution of healthcare "City clinical hospital 12", Saratov
  - State budget institution of healthcare of Yaroslavl region Regional clinical hospital, Yaroslavl
- Serbia (4):
  - Clinical Centre of Serbia, Clinic for Gastroenterology and Hepatology, Belgrade
  - Clinical Centre of Vojvodina, Clinic for Gastroenterology and Hepatology, Novi Sad
  - Clinical Centre of Vojvodina, Emergency Internal Medicine Division, Novi Sad
  - General Hospital Subotica, Subotica
- Slovakia (4):
  - Lama Medical Care s.r.o., Gastroenterologicko-Hepatologicke centrum Thalion, Bratislava
  - KM Management spol. s r.o., Nitra
  - Aura SA, s.r.o., Nové Mesto nad Váhom
  - Gastro I., s.r.o., Prešov
- South Africa (3):
  - Panorama Medi-Clinic, Cape Town, Western Cape
  - The Louis Leipoldt Medical Centre, Cape Town, Western Cape
  - Dr JP Wright, Claremont, Cape Town, Western Cape
- South Korea (9):
  - Hanyang University Guri Hospital, Clinical Laboratory, Guri-si, Gyeonggi-do
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do
  - Pusan National University Hospital, Busan
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Kyung Hee University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
- Spain (2):
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
- Taiwan (2):
  - Chung Shan Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- Ukraine (9):
  - Kyiv City Clinical Hospital #8,, Kiev, Ukraine
  - Regional Municipal Institution "Chernivtsi Regional Clinical Hospital", Chernivtsi
  - Regional Municipal Institution Chernivtsi Regional Clinical Hospital, Chernivtsi
  - State Institution Institute of Gastroenterology of the National Academy of Medical Sciences, Dnipropetrovsk
  - Municipal Healthcare Institution Kharkiv City Clinical Hospital #2, Proctology Department, Kharkiv
  - Municipal Institution "Odesa Regional Clinical Hospital", Odesa
  - Medical Clinical Research Center "Health Clinic" on the base of, Vinnytsia
  - Motor-Sich clinic, LLC, Zaporizhzhia
  - Minicipal Institution "City Hospital #7" Therapeutic Department,, Zaporizhzhia
- United Kingdom (4):
  - Department of Gastroenterology, Old Building, Bristol, England
  - St Mark's Hospital, Harrow, Middlesex
  - Norfolk and Norwich University Hospital, Norwich, Norfolk
  - Norfolk and Norwich University Hospital, Norwich

REFERENCES:
- [Derived] Panes J, D'Haens GR, Sands BE, Ng SC, Lawendy N, Kulisek N, Guo X, Wu J, Vranic I, Panaccione R, Vermeire S. Analysis of tofacitinib safety in ulcerative colitis from the completed global clinical developmental program up to 9.2 years of drug exposure. United European Gastroenterol J. 2024 Jul;12(6):793-801. doi: 10.1002/ueg2.12584. Epub 2024 May 22. PMID 38778549
- [Derived] Rubin DT, Torres J, Regueiro M, Reinisch W, Prideaux L, Kotze PG, Tan FH, Gardiner S, Mundayat R, Cadatal MJ, Ng SC. Association Between Smoking Status and the Efficacy and Safety of Tofacitinib in Patients with Ulcerative Colitis. Crohns Colitis 360. 2024 Jan 20;6(1):otae004. doi: 10.1093/crocol/otae004. eCollection 2024 Jan. PMID 38425446
- [Derived] Rubin DT, Salese L, Cohen M, Kotze PG, Woolcott JC, Su C, Mundayat R, Paulissen J, Torres J, Long MD. Presence of risk factors associated with colectomy among patients with ulcerative colitis: a post hoc analysis of data from the tofacitinib OCTAVE ulcerative colitis clinical program. Therap Adv Gastroenterol. 2023 Aug 7;16:17562848231189122. doi: 10.1177/17562848231189122. eCollection 2023. PMID 37560161
- [Derived] Schreiber S, Rubin DT, Ng SC, Peyrin-Biroulet L, Danese S, Modesto I, Guo X, Su C, Kwok KK, Jo H, Chen Y, Yndestad A, Reinisch W, Dubinsky MC. Major Adverse Cardiovascular Events by Baseline Cardiovascular Risk in Patients with Ulcerative Colitis Treated with Tofacitinib: Data from the OCTAVE Clinical Programme. J Crohns Colitis. 2023 Nov 24;17(11):1761-1770. doi: 10.1093/ecco-jcc/jjad104. PMID 37402275
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Lichtenstein GR, Cohen BL, Salese L, Modesto I, Wang W, Chan G, Ahmed HM, Su C, Peyrin-Biroulet L. Impact of Concomitant Corticosteroids on Tofacitinib Induction Efficacy and Infection Rates in Ulcerative Colitis. Dig Dis Sci. 2023 Jun;68(6):2624-2634. doi: 10.1007/s10620-022-07794-0. Epub 2023 Feb 4. PMID 36739367
- [Derived] Dubinsky MC, Armuzzi A, Gecse KB, Ullman T, Bushmakin AG, DiBonaventura M, Cappelleri JC, Connelly SB, Woolcott JC, Salese L. Improvements in Disease Activity Partially Mediate the Effect of Tofacitinib Treatment on Generic and Disease-Specific Health-Related Quality of Life in Patients with Ulcerative Colitis: Data from the OCTAVE Program. Dig Dis. 2023;41(4):604-614. doi: 10.1159/000528788. Epub 2023 Jan 5. PMID 36603566
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Sandborn WJ, Sands BE, Vermeire S, Leung Y, Guo X, Modesto I, Su C, Wang W, Panes J. Modified Mayo score versus Mayo score for evaluation of treatment efficacy in patients with ulcerative colitis: data from the tofacitinib OCTAVE program. Therap Adv Gastroenterol. 2022 Dec 5;15:17562848221136331. doi: 10.1177/17562848221136331. eCollection 2022. PMID 36506749
- [Derived] Lichtenstein GR, Bressler B, Francisconi C, Vermeire S, Lawendy N, Salese L, Sawyerr G, Shi H, Su C, Judd DT, Jones T, Loftus EV. Assessment of Safety and Efficacy of Tofacitinib, Stratified by Age, in Patients from the Ulcerative Colitis Clinical Program. Inflamm Bowel Dis. 2023 Jan 5;29(1):27-41. doi: 10.1093/ibd/izac084. PMID 36342120
- [Derived] Hudesman DP, Torres J, Salese L, Woolcott JC, Mundayat R, Su C, Mosli MH, Allegretti JR. Long-Term Improvement in the Patient-Reported Outcomes of Rectal Bleeding, Stool Frequency, and Health-Related Quality of Life with Tofacitinib in the Ulcerative Colitis OCTAVE Clinical Program. Patient. 2023 Mar;16(2):95-103. doi: 10.1007/s40271-022-00603-w. Epub 2022 Nov 7. PMID 36336750
- [Derived] Targownik L, Dubinsky MC, Steinwurz F, Bushmakin AG, Cappelleri JC, Tai E, Gardiner S, Hur P, Panes J. Disease Activity and Health-related Quality of Life Relationships with Work Productivity in Patients with Ulcerative Colitis in OCTAVE Induction 1 and 2 and OCTAVE Sustain. J Crohns Colitis. 2023 Apr 19;17(4):513-523. doi: 10.1093/ecco-jcc/jjac161. PMID 36271912
- [Derived] Sandborn WJ, D'Haens GR, Sands BE, Panaccione R, Ng SC, Lawendy N, Kulisek N, Modesto I, Guo X, Mundayat R, Su C, Vranic I, Panes J. Tofacitinib for the Treatment of Ulcerative Colitis: An Integrated Summary of up to 7.8 Years of Safety Data from the Global Clinical Programme. J Crohns Colitis. 2023 Apr 3;17(3):338-351. doi: 10.1093/ecco-jcc/jjac141. PMID 36124702
- [Derived] Loftus EV, Baumgart DC, Gecse K, Kinnucan JA, Connelly SB, Salese L, Su C, Kwok KK, Woolcott JC, Armuzzi A. Clostridium difficile Infection in Patients with Ulcerative Colitis Treated with Tofacitinib in the Ulcerative Colitis Program. Inflamm Bowel Dis. 2023 May 2;29(5):744-751. doi: 10.1093/ibd/izac139. PMID 35792493
- [Derived] Winthrop KL, Vermeire S, Long MD, Panes J, Ng SC, Kulisek N, Mundayat R, Lawendy N, Vranic I, Modesto I, Su C, Melmed GY. Long-term Risk of Herpes Zoster Infection in Patients With Ulcerative Colitis Receiving Tofacitinib. Inflamm Bowel Dis. 2023 Jan 5;29(1):85-96. doi: 10.1093/ibd/izac063. PMID 35648151
- [Derived] Mukherjee A, Tsuchiwata S, Nicholas T, Cook JA, Modesto I, Su C, D'Haens GR, Sandborn WJ. Exposure-Response Characterization of Tofacitinib Efficacy in Moderate to Severe Ulcerative Colitis: Results From Phase II and Phase III Induction and Maintenance Studies. Clin Pharmacol Ther. 2022 Jul;112(1):90-100. doi: 10.1002/cpt.2601. Epub 2022 Apr 27. PMID 35380740
- [Derived] Dubinsky MC, Magro F, Steinwurz F, Hudesman DP, Kinnucan JA, Ungaro RC, Neurath MF, Kulisek N, Paulissen J, Su C, Ponce de Leon D, Regueiro M. Association of C-reactive Protein and Partial Mayo Score With Response to Tofacitinib Induction Therapy: Results From the Ulcerative Colitis Clinical Program. Inflamm Bowel Dis. 2023 Jan 5;29(1):51-61. doi: 10.1093/ibd/izac061. PMID 35380664
- [Derived] Feagan BG, Khanna R, Sandborn WJ, Vermeire S, Reinisch W, Su C, Salese L, Fan H, Paulissen J, Woodworth DA, Niezychowski W, Sands BE. Agreement between local and central reading of endoscopic disease activity in ulcerative colitis: results from the tofacitinib OCTAVE trials. Aliment Pharmacol Ther. 2021 Dec;54(11-12):1442-1453. doi: 10.1111/apt.16626. Epub 2021 Oct 6. PMID 34614208
- [Derived] Farraye FA, Qazi T, Kotze PG, Moore GT, Mundayat R, Lawendy N, Sharma PP, Judd DT. The impact of body mass index on efficacy and safety in the tofacitinib OCTAVE ulcerative colitis clinical programme. Aliment Pharmacol Ther. 2021 Aug;54(4):429-440. doi: 10.1111/apt.16439. Epub 2021 Jun 24. PMID 34165201
- [Derived] Rubin DT, Reinisch W, Greuter T, Kotze PG, Pinheiro M, Mundayat R, Maller E, Fellmann M, Lawendy N, Modesto I, Vavricka SR, Lichtenstein GR. Extraintestinal manifestations at baseline, and the effect of tofacitinib, in patients with moderate to severe ulcerative colitis. Therap Adv Gastroenterol. 2021 May 16;14:17562848211005708. doi: 10.1177/17562848211005708. eCollection 2021. PMID 34035832
- [Derived] Sandborn WJ, Peyrin-Biroulet L, Sharara AI, Su C, Modesto I, Mundayat R, Gunay LM, Salese L, Sands BE. Efficacy and Safety of Tofacitinib in Ulcerative Colitis Based on Prior Tumor Necrosis Factor Inhibitor Failure Status. Clin Gastroenterol Hepatol. 2022 Mar;20(3):591-601.e8. doi: 10.1016/j.cgh.2021.02.043. Epub 2021 Mar 6. PMID 33684552
- [Derived] Vong C, Martin SW, Deng C, Xie R, Ito K, Su C, Sandborn WJ, Mukherjee A. Population Pharmacokinetics of Tofacitinib in Patients With Moderate to Severe Ulcerative Colitis. Clin Pharmacol Drug Dev. 2021 Mar;10(3):229-240. doi: 10.1002/cpdd.899. Epub 2021 Jan 29. PMID 33513294
- [Derived] Curtis JR, Regueiro M, Yun H, Su C, DiBonaventura M, Lawendy N, Nduaka CI, Koram N, Cappelleri JC, Chan G, Modesto I, Lichtenstein GR. Tofacitinib Treatment Safety in Moderate to Severe Ulcerative Colitis: Comparison of Observational Population Cohort Data From the IBM MarketScan(R) Administrative Claims Database With Tofacitinib Trial Data. Inflamm Bowel Dis. 2021 Aug 19;27(9):1394-1408. doi: 10.1093/ibd/izaa289. PMID 33324993
- [Derived] Sandborn WJ, Peyrin-Biroulet L, Quirk D, Wang W, Nduaka CI, Mukherjee A, Su C, Sands BE. Efficacy and Safety of Extended Induction With Tofacitinib for the Treatment of Ulcerative Colitis. Clin Gastroenterol Hepatol. 2022 Aug;20(8):1821-1830.e3. doi: 10.1016/j.cgh.2020.10.038. Epub 2020 Oct 27. PMID 33127596
- [Derived] Sands BE, Colombel JF, Ha C, Farnier M, Armuzzi A, Quirk D, Friedman GS, Kwok K, Salese L, Su C, Taub PR. Lipid Profiles in Patients With Ulcerative Colitis Receiving Tofacitinib-Implications for Cardiovascular Risk and Patient Management. Inflamm Bowel Dis. 2021 May 17;27(6):797-808. doi: 10.1093/ibd/izaa227. PMID 32870265
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Dubinsky MC, DiBonaventura M, Fan H, Bushmakin AG, Cappelleri JC, Maller E, Thorpe AJ, Salese L, Panes J. Tofacitinib in Patients with Ulcerative Colitis: Inflammatory Bowel Disease Questionnaire Items in Phase 3 Randomized Controlled Induction Studies. Inflamm Bowel Dis. 2021 Jun 15;27(7):983-993. doi: 10.1093/ibd/izaa193. PMID 32794567
- [Derived] Lichtenstein GR, Rogler G, Ciorba MA, Su C, Chan G, Pedersen RD, Lawendy N, Quirk D, Nduaka CI, Thorpe AJ, Panes J. Tofacitinib, an Oral Janus Kinase Inhibitor: Analysis of Malignancy (Excluding Nonmelanoma Skin Cancer) Events Across the Ulcerative Colitis Clinical Program. Inflamm Bowel Dis. 2021 May 17;27(6):816-825. doi: 10.1093/ibd/izaa199. PMID 32766762
- [Derived] Sandborn WJ, Panes J, Sands BE, Reinisch W, Su C, Lawendy N, Koram N, Fan H, Jones TV, Modesto I, Quirk D, Danese S. Venous thromboembolic events in the tofacitinib ulcerative colitis clinical development programme. Aliment Pharmacol Ther. 2019 Nov;50(10):1068-1076. doi: 10.1111/apt.15514. Epub 2019 Oct 9. PMID 31599001
- [Derived] Sands BE, Taub PR, Armuzzi A, Friedman GS, Moscariello M, Lawendy N, Pedersen RD, Chan G, Nduaka CI, Quirk D, Salese L, Su C, Feagan BG. Tofacitinib Treatment Is Associated With Modest and Reversible Increases in Serum Lipids in Patients With Ulcerative Colitis. Clin Gastroenterol Hepatol. 2020 Jan;18(1):123-132.e3. doi: 10.1016/j.cgh.2019.04.059. Epub 2019 May 8. PMID 31077827
- [Derived] Sandborn WJ, Panes J, D'Haens GR, Sands BE, Su C, Moscariello M, Jones T, Pedersen R, Friedman GS, Lawendy N, Chan G. Safety of Tofacitinib for Treatment of Ulcerative Colitis, Based on 4.4 Years of Data From Global Clinical Trials. Clin Gastroenterol Hepatol. 2019 Jul;17(8):1541-1550. doi: 10.1016/j.cgh.2018.11.035. Epub 2018 Nov 23. PMID 30476584
- [Derived] Hanauer S, Panaccione R, Danese S, Cheifetz A, Reinisch W, Higgins PDR, Woodworth DA, Zhang H, Friedman GS, Lawendy N, Quirk D, Nduaka CI, Su C. Tofacitinib Induction Therapy Reduces Symptoms Within 3 Days for Patients With Ulcerative Colitis. Clin Gastroenterol Hepatol. 2019 Jan;17(1):139-147. doi: 10.1016/j.cgh.2018.07.009. Epub 2018 Sep 10. PMID 30012431
- [Derived] Winthrop KL, Melmed GY, Vermeire S, Long MD, Chan G, Pedersen RD, Lawendy N, Thorpe AJ, Nduaka CI, Su C. Herpes Zoster Infection in Patients With Ulcerative Colitis Receiving Tofacitinib. Inflamm Bowel Dis. 2018 Sep 15;24(10):2258-2265. doi: 10.1093/ibd/izy131. PMID 29850873
- [Derived] Motoya S, Watanabe M, Kim HJ, Kim YH, Han DS, Yuasa H, Tabira J, Isogawa N, Arai S, Kawaguchi I, Hibi T. Tofacitinib induction and maintenance therapy in East Asian patients with active ulcerative colitis: subgroup analyses from three phase 3 multinational studies. Intest Res. 2018 Apr;16(2):233-245. doi: 10.5217/ir.2018.16.2.233. Epub 2018 Apr 30. PMID 29743836
- [Derived] Panes J, Vermeire S, Lindsay JO, Sands BE, Su C, Friedman G, Zhang H, Yarlas A, Bayliss M, Maher S, Cappelleri JC, Bushmakin AG, Rubin DT. Tofacitinib in Patients with Ulcerative Colitis: Health-Related Quality of Life in Phase 3 Randomised Controlled Induction and Maintenance Studies. J Crohns Colitis. 2018 Jan 24;12(2):145-156. doi: 10.1093/ecco-jcc/jjx133. PMID 29028981
- [Derived] Sandborn WJ, Su C, Sands BE, D'Haens GR, Vermeire S, Schreiber S, Danese S, Feagan BG, Reinisch W, Niezychowski W, Friedman G, Lawendy N, Yu D, Woodworth D, Mukherjee A, Zhang H, Healey P, Panes J; OCTAVE Induction 1, OCTAVE Induction 2, and OCTAVE Sustain Investigators. Tofacitinib as Induction and Maintenance Therapy for Ulcerative Colitis. N Engl J Med. 2017 May 4;376(18):1723-1736. doi: 10.1056/NEJMoa1606910. PMID 28467869
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921095&StudyName=A%20Study%20To%20Evaluate%20Both%20The%20Efficacy%20and%20Safety%20Profile%20of%20CP-690%2C550%20In%20Patients%20With%20Moderately%20to%20Severely%20Active%20Ulcerative%20Col

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to tofacitinib 10 milligram (mg) or placebo twice a day (BID)(4:1 ratio) after Protocol Amendment 2, which removed tofacitinib 15 mg BID. Due to low participant numbers, tofacitinib 15 mg BID was excluded from efficacy analyses, but was included in participant flow, baseline characteristics and adverse events analyses.
Groups:
- Tofacitinib 10 mg BID: Participants received tofacitinib 10 mg tablets, orally, BID for 9 weeks of double blind treatment period.
- Tofacitinib 15 mg BID: Participants received tofacitinib 15 mg tablets, orally, BID for 9 weeks of double blind treatment period.
- Placebo BID: Participants received tofacitinib-matched placebo tablets, orally, BID for 9 weeks of double blind treatment period.
Period: Overall Study
Arm/Group | Tofacitinib 10 mg BID | Tofacitinib 15 mg BID | Placebo BID
Started | 429 | 6 | 112
Completed | 397 | 5 | 97
Not Completed | 32 | 1 | 15
Not completed — Other | 1 | 0 | 0
Not completed — Protocol Violation | 5 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 2
Not completed — Adverse Event | 7 | 0 | 2
Not completed — Insufficient Clinical Response | 17 | 0 | 11

BASELINE CHARACTERISTICS:
Population: The safety analysis set consists of all randomized participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tofacitinib 10 mg BID | Tofacitinib 15 mg BID | Placebo BID | Total
Number analyzed (Participants) | 429 | 6 | 112 | 547
Age, Customized [Number; unit: participants]
  18 to 44 Years | 265 | 5 | 72 | 342
  45 to 64 Years | 139 | 1 | 35 | 175
  Greater Than or Equal to (>=) 65 Years | 25 | 0 | 5 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 170 | 3 | 57 | 230
  Male | 259 | 3 | 55 | 317

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Remission at Week 8
Description: Remission in participants was defined by a total Mayo score of 2 points or lower, with no individual subscore exceeding 1 point and a rectal bleeding subscore of 0. Mayo score is an instrument designed to measure disease activity of Ulcerative Colitis . It consisted of 4 subscores: stool frequency, rectal bleeding, findings of centrally read flexible proctosigmoidoscopy and physician global assessment (PGA), each graded from 0 to 3 with higher scores indicating more severe disease. These scores were summed up to give a total score range of 0 to 12; where higher score indicating more severe disease.
Time Frame: Week 8
Population: Full analysis set included all participants who were randomly assigned to either tofacitinib 10 mg BID or placebo BID.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 429 | 112
percentage of participants | 16.6 | 3.6
Statistical Analysis 1: Comparison: Tofacitinib 10 mg BID vs Placebo BID; P-value based on Cochran-Mantel Haenszel (CMH) chi-square test stratified by prior treatment with anti-tumor necrosis factor (TNF), steroid use at baseline and geographic region. Percentage difference and its 95% CI was based on normal approximation for the difference in binomial proportions. Missing data were imputed using non-responder imputation (NRI); Test type: Superiority or Other; p = 0.0005, CMH Chi-square Test; Percentage difference = 13.0, 95% CI 2-sided [8.1 to 17.9]

2. Secondary Outcome: Percentage of Participants Achieving Mucosal Healing at Week 8
Description: Mucosal healing in participants was defined by Mayo endoscopic subscore of 0 or 1. The Mayo endoscopic subscore consisted of the findings of centrally read flexible proctosigmoidoscopy, graded from 0 to 3 with higher scores indicating more severe disease.
Time Frame: Week 8
Population: Full analysis set included all participants who were randomly assigned to either tofacitinib 10 mg BID or placebo BID.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 429 | 112
percentage of participants | 28.4 | 11.6
Statistical Analysis 1: Comparison: Tofacitinib 10 mg BID vs Placebo BID; P-value was based on CMH chi-square test stratified by prior treatment with anti-TNF, steroid use at baseline and geographic region. Percentage difference and its 95% CI was based on normal approximation for the difference in binomial proportions. Missing data were imputed using NRI; Test type: Superiority or Other; p = 0.0002, CMH Chi-square Test; Percentage difference = 16.8, 95% CI 2-sided [9.5 to 24.1]

3. Secondary Outcome: Percentage of Participants Achieving Clinical Response at Week 8
Description: Clinical response in participants was defined by a decrease from baseline in Mayo score of at least 3 points and at least 30 percent, with an accompanying decrease in the rectal bleeding sub score of at least 1 point or an absolute rectal bleeding sub score of 0 or 1. Mayo score is an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of flexible centrally read proctosigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating more severe disease. These scores were summed up to give a total score range of 0 to 12; where higher score indicating more severe disease.
Time Frame: Week 8
Population: Full analysis set included all participants who were randomly assigned to either tofacitinib 10 mg BID or placebo BID.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 429 | 112
percentage of participants | 55.0 | 28.6
Statistical Analysis 1: Comparison: Tofacitinib 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, CMH Chi-square Test; Percentage difference = 26.4, 95% CI 2-sided [16.8 to 36.0]

4. Secondary Outcome: Percentage of Participants With Endoscopic Remission at Week 8
Description: Endoscopic remission in participants was defined by Mayo endoscopic subscore of 0. The Mayo endoscopic subscore consisted of the findings of centrally read flexible proctosigmoidoscopy, graded from 0 to 3 with higher scores indicating more severe disease.
Time Frame: Week 8
Population: Full analysis set included all participants who were randomly assigned to either tofacitinib 10 mg BID or placebo BID.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 429 | 112
percentage of participants | 7.0 | 1.8
Statistical Analysis 1: Comparison: Tofacitinib 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0425, CMH Chi-square Test; Percentage difference = 5.2, 95% CI 2-sided [1.8 to 8.6]

5. Secondary Outcome: Percentage of Participants With Clinical Remission at Week 8
Description: Clinical remission in participants was defined by a total Mayo score of 2 points or lower, with no individual subscore exceeding 1 point. Mayo score is an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of flexible centrally read proctosigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating more severe disease. These scores were summed up to give a total score range of 0 to 12; where higher score indicating more severe disease.
Time Frame: Week 8
Population: Full analysis set included all participants who were randomly assigned to either tofacitinib 10 mg BID or placebo BID.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 429 | 112
percentage of participants | 16.8 | 3.6
Statistical Analysis 1: Comparison: Tofacitinib 10 mg BID vs Placebo BID; P-value was based on CMH chi-square test stratified by prior treatment with anti-TNF, steroid use at baseline and geographic region. Difference in its percentage and its 95% CI was based on normal approximation for the difference in binomial proportions. Missing data were imputed using NRI; Test type: Superiority or Other; p = 0.0004, CMH Chi-square Test; Difference in percentage = 13.2, 95% CI 2-sided [8.3 to 18.1]

6. Secondary Outcome: Percentage of Participants With Symptomatic Remission at Week 8
Description: Symptomatic remission was defined by a total Mayo score of 2 points or lower, with no individual subscore exceeding 1 point, and 0 subscore for both rectal bleeding and stool frequency. Mayo score is an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of flexible centrally read proctosigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating more severe disease. These scores were summed up to give a total score range of 0 to 12; where higher score indicating more severe disease.
Time Frame: Week 8
Population: Full analysis set included all participants who were randomly assigned to either tofacitinib 10 mg BID or placebo BID.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 429 | 112
percentage of participants | 10.7 | 2.7
Statistical Analysis 1: Comparison: Tofacitinib 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0090, CMH Chi-square Test; Percentage difference = 8.0, 95% CI 2-sided [3.9 to 12.2]

7. Secondary Outcome: Percentage of Participants With Deep Remission at Week 8
Description: Deep remission in participants was defined by a total Mayo score of 2 points or lower, with no individual subscore exceeding 1 point and 0 subscore for both rectal bleeding and endoscopic subscores. Mayo score is an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of flexible centrally read proctosigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating more severe disease. These scores were summed up to give a total score range of 0 to 12; where higher score indicating more severe disease.
Time Frame: Week 8
Population: Full analysis set included all participants who were randomly assigned to either tofacitinib 10 mg BID or placebo BID.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 429 | 112
percentage of participants | 5.1 | 1.8
Statistical Analysis 1: Comparison: Tofacitinib 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1408, CMH Chi-square Test; Percentage difference = 3.3, 95% CI 2-sided [0.1 to 6.6]

8. Secondary Outcome: Partial Mayo Scores
Description: A partial mayo score (mayo score without endoscopy) ranges from 0 (normal or inactive disease) to 9 (severe disease) and calculated as the sum of 3 subscores (stool frequency, rectal bleeding and PGA) and each grading from 0 to 3 with higher scores indicating more severe disease.
Time Frame: Baseline, Weeks 2, 4, 8
Population: Full analysis set included all participants who were randomly assigned to either tofacitinib 10 mg BID or placebo BID. Here, 'n' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 429 | 112
units on a scale
  Baseline (n= 428, 112 ) | 6.4 (1.3) | 6.4 (1.2)
  Week 2 (n= 419, 107 ) | 4.4 (2.2) | 5.4 (1.7)
  Week 4 (n= 412, 102 ) | 3.7 (2.3) | 4.8 (2.0)
  Week 8 (n= 401, 98 ) | 3.3 (2.3) | 4.5 (2.1)

9. Secondary Outcome: Change From Baseline in Partial Mayo Scores at Weeks 2, 4 and 8
Description: Change in Partial Mayo scores at Weeks 2, 4, 8 relative to baseline were reported. A Partial Mayo Score (Mayo score without endoscopy) ranges from 0 (normal or inactive disease) to 9 (severe disease) and calculated as the sum of 3 subscores (stool frequency, rectal bleeding and PGA) with each graded from 0 to 3 with higher scores indicating more severe disease.
Time Frame: Baseline, Weeks 2, 4, 8
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 429 | 112
units on a scale
  Change at Week 2 (n= 418, 107 ) | -2.0 (0.1) | -1.0 (0.2)
  Change at Week 4 (n= 411, 102 ) | -2.7 (0.1) | -1.5 (0.2)
  Change at Week 8 (n= 400, 98 ) | -3.0 (0.1) | -1.7 (0.2)
Statistical Analysis 1: Comparison: Tofacitinib 10 mg BID vs Placebo BID; At Week 2: The change from baseline was analyzed using mixed effect model with treatment group, prior treatment with antiTNF, steroid use at baseline, geographic region, visit and visit by treatment group all as fixed effects, and subjects as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Least square mean difference = -1.0, 95% CI 2-sided [-1.4 to -0.6], Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo BID; At Week 4: The change from baseline was analyzed using mixed effect model with treatment group, prior treatment with antiTNF, steroid use at baseline, geographic region, visit and visit by treatment group all as fixed effects, and subjects as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Least square mean difference = -1.2, 95% CI 2-sided [-1.6 to -0.7], Standard Error of Mean 0.2
Statistical Analysis 3: Comparison: Tofacitinib 10 mg BID vs Placebo BID; At Week 8: The change from baseline was analyzed using mixed effect model with treatment group, prior treatment with antiTNF, steroid use at baseline, geographic region, visit and visit by treatment group all as fixed effects, and subjects as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Least square mean difference = -1.3, 95% CI 2-sided [-1.7 to -0.9], Standard Error of Mean 0.2

10. Secondary Outcome: Change From Baseline in Total Mayo Score at Week 8
Description: Change in total Mayo scores at Week 8 relative to Baseline was reported. Mayo score is an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of flexible centrally read proctosigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating more severe disease. These scores were summed up to give a total score range of 0 to 12; where higher score indicating more severe disease.
Time Frame: Baseline, Week 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 429 | 112
units on a scale
  Baseline (n=428,112) | 9.0 (1.5) | 8.9 (1.5)
  Change at Week 8 (n=396,98) | -3.7 (2.8) | -2.0 (2.4)
Statistical Analysis 1: Comparison: Tofacitinib 10 mg BID vs Placebo BID; The change from baseline at Week 8 was analyzed using an analysis of covariance (ANCOVA) model with treatment group, prior treatment with anti-TNF, steroid use at baseline and geographic region as factors and baseline as a covariate based on the observed-case data; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Square Mean Difference = -1.6, 95% CI 2-sided [-2.2 to -1.0], Standard Error of Mean 0.3

ADVERSE EVENTS:
Time Frame: Baseline up to Day 98
Description: The same event may appear as both an adverse event (AE) and an serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non serious event during the study.
Arm/Group | Tofacitinib 10 mg BID | Tofacitinib 15 mg BID | Placebo BID
Serious Adverse Events (participants affected / at risk) | 18/429 | 0/6 | 9/112
Other Adverse Events (participants affected / at risk) | 68/429 | 4/6 | 20/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib 10 mg BID (N=429) | Tofacitinib 15 mg BID (N=6) | Placebo BID (N=112)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 8 | 0 | 4
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib 10 mg BID (N=429) | Tofacitinib 15 mg BID (N=6) | Placebo BID (N=112)
Anaemia (Blood and lymphatic system disorders) | 11 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 7 | 0 | 6
Abdominal pain upper (Gastrointestinal disorders) | 7 | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Urine analysis abnormal (Investigations) | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 0 | 6
Headache (Nervous system disorders) | 33 | 0 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.